CLINICAL TRIAL: NCT00582426
Title: LARCID: Evaluation of Octreotide LAR in Prevention of Chemotherapy-induced Diarrhea
Brief Title: Evaluation of Octreotide LAR in Prevention of Chemotherapy-induced Diarrhea
Acronym: LARCID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSMS995AIC04
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Chemotherapy-induced Diarrhea
Keywords: Colorectal cancer; diarrhea; drug therapy; octreotide; fluorouracil; irinotecan; capecitabine; prevention
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea

ARMS (2):
- Octreotide Long Acting Release (Experimental): Prevention of Chemotherapy Induced Diarrhea (CID)
  Interventions: Drug: Octreotide Long Acting Release
- Standard Treatment (Other): Physician treatment of choice for chemotherapy induced diarrhea other than Octreotide LAR.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Drug: Octreotide Long Acting Release — Patients will receive the first dose of Octreotide LAR (30 mg) at chemotherapy initiation, in addition to a minimum of two more identical monthly doses of Octreotide LAR (with an interval of 28 days between them), until first-line chemotherapy is discontinued or for a maximum of six doses of Octreotide LAR, whichever occurs first.
  Other Names: Octreotide LAR; Sandostatin LAR
  Arms: Octreotide Long Acting Release
Other: Standard Treatment — Physician treatment of choice for chemotherapy induced diarrhea other than Octreotide LAR.
  Arms: Standard Treatment

SUMMARY:
This study will evaluate the efficacy of Octreotide LAR in preventing chemotherapy-induced diarrhea (with regimens that contain 5 fluorouracil, irinotecan and capecitabine)in patients with colorectal cancer.

DETAILED DESCRIPTION:
Eligible patients will have a diagnosis of colorectal cancer, and will be candidates to adjuvant chemotherapy or first-line chemotherapy for metastatic disease with a regimen containing fluorouracil, capecitabine and/or irinotecan. Eligible chemotherapy regimens include Irinotecan, Leucovorin (folinic acid), and Fluorouracil(IFL), Leucovorin, Fluorouracil, and Irinotecan (FOLFIRI), combinations of Irinotecan and Capecitabine, the Roswell Park regimen and the Mayo Clinic regimen, all of them without or with Oxaliplatin, Bevacizumab or Cetuximab. Patients receiving Erlotinib, or other Tyrosine-kinase, Epidermal Growth Factor Receptor (EGFR)-inhibitors, will not be eligible.

The acute treatment for diarrhea will be left to physician's discretion in both groups. Patients in the control arm will be treated without Octreotide LAR. Patients in the experimental arm will receive the first dose of Octreotide LAR (30 mg) at chemotherapy initiation, in addition to a minimum of two more identical monthly doses of Octreotide LAR (with an interval of 28 days between them), until chemotherapy is discontinued or for a maximum of six doses of Octreotide LAR, whichever occurs first. Patient evaluation will be done at each cycle for efficacy and toxicity.

ELIGIBILITY:
Inclusion criteria:

1. Providing a written informed consent
2. Age between 18 and 80 years;
3. Histological diagnosis of colorectal cancer, presence of metastatic disease and no prior systemic therapy for metastatic disease (prior adjuvant therapy will be allowed if completed 6 months or longer before inclusion in the study);
4. Indication of treatment, according to the judgment of the investigator, with a chemotherapy regimen containing either 5-FU, capecitabine, or irinotecan; any such regimen may also include oxaliplatin, bevacizumab, or cetuximab;
5. A performance status of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale
6. Adequate organ function and lab values within specific ranges
7. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration;
8. Fertile patients (male or female) must agree to use an acceptable method of contraception to avoid pregnancy for the duration of the study and for 3 months after study termination;
9. No prior use of octreotide in any formulation.

Exclusion criteria:

1. Use of concomitant antineoplastic treatments, other than regimens containing either 5-FU, capecitabine, or irinotecan with or without oxaliplatin, bevacizumab, or cetuximab;
2. Previous or concomitant need for radiotherapy to the abdomen or pelvis;
3. Indication of treatment, according to the judgment of the investigator, with erlotinib, gefitinib, panitumumab, or other EGFR-inhibitors other than cetuximab;
4. A second malignancy (except in situ carcinoma of the cervix, in situ carcinoma of the bladder, adequately treated basal-cell or squamous-cell carcinoma of the skin, or another malignancy treated more than 5 years prior to enrollment and without recurrence);
5. Any type of condition leading to chronic diarrhea, including, but not limited to inflammatory bowel disease (e.g., ulcerative colitis and Crohn's disease), chronic diarrhea of presumed or confirmed infectious origin, and irritable bowel syndrome;
6. Active or uncontrolled concurrent medical condition, including, but not limited to, unstable angina, congestive heart failure, coronary artery disease, hypertension, diabetes mellitus, and hyper- or hypothyroidism;
7. Active and ongoing systemic infection;
8. Serious uncontrolled psychiatric illness;
9. Ongoing pregnancy or lactation;
10. Female patients who are pregnant or lactating, or are of childbearing potential and would not practice a medically acceptable method for birth control;
11. Lesions that have been irradiated cannot be included as sites of measurable disease. If the only measurable lesion was previously irradiated the patient cannot be included;
12. Use of any investigational agent within 30 days prior to enrollment in the study or foreseen use of an investigational agent during the study;
13. History of chronic (≥ 30 nonconsecutive days) use of laxatives;
14. Concurrent use of antidiarrheal agents;
15. Inability to comply with the study protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Brazil (11):
  - Biocâncer, Belo Horizonte
  - CEPON-Centro de Pesquisas Oncologicas, Florianópolis
  - Hospital Sao Lucas- Faculdade de Medicina da PUCRS, Porto Alegre
  - Clínica AMO, Salvador
  - Nucleo de Oncologia da Bahia, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - Hosital Alemão Oswaldo Cruz, São Paulo
  - Hospital A C Camargo/ Fundação Antonio Prudente, São Paulo
  - Hospital das Clínicas - FMUSP, São Paulo
  - Instituto Arnaldo Vieira de Carvalho - IAVC, São Paulo
  - UNIFESP, São Paulo

REFERENCES:
- [Derived] Hoff PM, Saragiotto DF, Barrios CH, del Giglio A, Coutinho AK, Andrade AC, Dutra C, Forones NM, Correa M, Portella Mdo S, Passos VQ, Chinen RN, van Eyll B. Randomized phase III trial exploring the use of long-acting release octreotide in the prevention of chemotherapy-induced diarrhea in patients with colorectal cancer: the LARCID trial. J Clin Oncol. 2014 Apr 1;32(10):1006-11. doi: 10.1200/JCO.2013.50.8077. Epub 2014 Feb 10. PMID 24516038

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide Long Acting Release: Octreotide LAR 30 mg, for intramuscular injection every 28 days for 6 months beginning with the first course of chemotherapy.
Period: Overall Study
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Started | 68 (Patient in both arms belongs to "started" indicates safety and intent to treat (ITT) populations.) | 71
Completed | 48 | 58
Not Completed | 20 | 13
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Protocol Violation | 6 | 2
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Disease Progression | 2 | 2
Not completed — Use of illicit drugs | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide Long Acting Release | Standard Treatment | Total
Number analyzed (Participants) | 68 | 71 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (12.8) | 55.5 (11.4) | 55.85 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Developing Diarrhea (Grade 1 to 4)
Description: The percentage of patients developing diarrhea (incidence of grade 1 to 4) during treatment, considering only the worst grade of diarrhea for each patient. Diarrhea was graded according to Common Toxicity Criteria where Grade 0=None, 1 = Increase of <4 stools/day over pretreatment, Grade 2 = Increase of 4-6 stools/day, or nocturnal stools, Grade 3 = Increase of ≥7 stools/day or incontinence; or need for parenteral support for dehydration and Grade 4= Physiologic consequences requiring intensive care; or hemodynamic collapse.
Time Frame: 6 month overall
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer. 1 patient from the "Octreotide Long Acting Release" Arm discontinued due to exclusion criteria after visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 67 | 71
Percentage of Participants | 76.1 [64.7 to 84.7] | 78.9 [68 to 86.8]

2. Secondary Outcome: Number of Episodes of Diarrhea by Patient
Description: Number of episodes of diarrhea is evaluated by patient diaries recorded on a daily basis.
Time Frame: 6 months overall
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer. Patients with observations during overall treatment period were included in this analysis.
Measure: Mean (Standard Deviation); unit: Episodes/patients/day
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 51 | 56
Episodes/patients/day | 21.6 (24.3) | 20.4 (19.6)

3. Secondary Outcome: Number of Episodes of Diarrhea by Patient by Cycle
Description: Mean number of episodes of diarrhea is evaluated by patient diaries recorded by cycle. (cycle 1 to cycle 7.)
Time Frame: at each cycle (28 days per cycle)
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer. "n" indicates patients with observations during each cycle.
Measure: Mean (Standard Deviation); unit: Episodes/patient/cycle
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 51 | 56
Episodes/patient/cycle
  Cycle 1 (n=20, 18) | 2.6 (2.2) | 2.2 (2)
  Cycle 2 (n=36,38) | 8.2 (6.8) | 5.9 (6.2)
  Cycle 3 (n=33,39) | 6.9 (7.8) | 6.7 (6.5)
  Cycle 4 (n=24, 27) | 8.6 (7.1) | 7.1 (7.1)
  Cycle 5 (n=20,29) | 8.1 (7.1) | 7 (8.8)
  Cycle 6 (n=22, 22) | 6.1 (6.9) | 5.8 (5.3)
  Cycle 7 (n= 16, 20) | 4.8 (6.3) | 6.6 (6.4)

4. Secondary Outcome: Percentage of Patients by Grade of Diarrhea
Description: Grade (severity) of episodes of diarrhea is evaluated by patient diaries recorded on a daily basis by considering only worse grade of diarrhea for each patient. Diarrhea was graded according to Common Toxicity Criteria where Grade 0 = None, 1 = Increase of <4 stools/day over pretreatment, Grade 2 = Increase of 4-6 stools/day, or nocturnal stools, Grade 3 = Increase of ≥7 stools/day or incontinence; or need for parenteral support for dehydration and Grade 4= Physiologic consequences requiring intensive care; or hemodynamic collapse.
Time Frame: 6 months overall
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 51 | 56
Percentage of Participants
  Grade 1 | 41.2 | 26.8
  Grade 2 | 25.5 | 51.8
  Grade 3 | 33.3 | 21.4
  Grade 4 | 0 | 0

5. Secondary Outcome: Percentage of Episodes by Grade
Description: Grade (severity)of episodes of diarrhea is evaluated by patient diaries recorded on a daily basis by considering only worse grade of diarrhea for each patient. Diarrhea was graded according to Common Toxicity Criteria where Grade 1 = Increase of <4 stools/day over pretreatment, Grade 2 = Increase of 4-6 stools/day, or nocturnal stools, Grade 3 = Increase of ≥7 stools/day or incontinence;or need for parenteral support for dehydration and Grade 4= Physiologic consequences requiring intensive care; or hemodynamic collapse.
Time Frame: 6 months overall
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer.
Measure: Number; unit: Percentage of Episodes
Units Other Than Participants: Episodes of Diarrhea
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 68 | 71
Number analyzed (Episodes of Diarrhea) | 257 | 272
Percentage of Episodes
  Grade 1 | 65.4 | 66.9
  Grade 2 | 23.3 | 27.2
  Grade 3 | 11.3 | 5.9
  Grade 4 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Need Chemotherapy Dose Reduction Due to Diarrhea
Description: For patient, chemotherapy dose reduction due to diarrhea as counted each time it occurred. Chemotherapy dose reduction because of other adverse events related to chemotherapy was not considered.
Time Frame: 6 months overall
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer. 1 patient discontinued from the Octreotide LAR arm due to exclusion criteria after visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 67 | 71
Percentage of participants | 26.9 [17.7 to 38.5] | 11.3 [5.8 to 20.7]

7. Secondary Outcome: Percentage of Participants Who Need Opioids for Control of Diarrhea
Time Frame: 6 months overall
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 67 | 71
Percentage of Participants | 1.5 [0.3 to 8.0] | 1.4 [0.2 to 7.6]

8. Secondary Outcome: Percentage of Patients Hospitalized Due to Diarrhea
Time Frame: 6 months overall
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 67 | 71
Percentage of patients | 6 | 4.2

9. Secondary Outcome: Percentage of Participants Who Need Intravenous Hydration for Control of Diarrhea
Time Frame: 6 months overall
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 67 | 71
Percentage of Participants | 4.5 [1.5 to 12.4] | 7.0 [3.0 to 15.4]

10. Secondary Outcome: Percentage of Participants With Complete or Partial Response at Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Lesions that can be accurately measured in at least one dimension (longest diameter (LD) to be recorded) as > 20 mm with conventional techniques (CT, MRI) or as > 10 mm with spiral CT scan. All measurable lesions up to maximum of 5 lesions per organ and 10 lesions in total representative of all involved organs should be identified as target lesions and recorded and measured at baseline. Complete Response is defined as Disappearance of all target lesions. Partial Response is defined at least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD.
Time Frame: Day 56, Day 84, Day 112, Day 140, Day 168
Population: ITT population includes all registered patients. Also considered in the intent to treat population are patients withdrawn prematurely from the study due to treatment interruption for a period of 28 consecutive days or longer. "N" in each category indicates the number of patients analyzed with observations at that timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 68 | 71
Percentage of Participants
  Day 56 (N=11,2) | 45.5 [21.3 to 72.0] | 0.0 [0.0 to 65.8]
  Day 84 (N=5,3) | 60.0 [23.1 to 88.2] | 100 [43.8 to 100]
  Day 112 (N=1,1) | 100 [20.7 to 100] | 0.0 [0.0 to 79.3]
  Day 140 (N=9,1) | 44.4 [18.9 to 73.3] | 100 [20.7 to 100]
  Day 168 (N=2,1) | 100 [34.2 to 100] | 100 [20.7 to 100]

11. Secondary Outcome: Change From Baseline in Quality of Life Measured by the Functional Assessment of Chronic Illness Therapy-Diarrhea (FACIT-D)
Description: Quality of life (QoL) is evaluated using FACIT-D scale. FACIT-D is composed of 38 items, whose responses range from 0 to 4. The total FACIT-D score may range from 0 to 152. The 38 items compose five subscales, each evaluating a different component of the (QOL). For calculating the subscale score, some items are computed in a reverse fashion, so that higher FACIT-D scores indicate a better (QoL). Descriptive statistics (mean, standard deviation, median, minimum and maximum) are used to summarize FACIT-D scores (total and subscales) by study group at each time point.
Time Frame: Baseline to Day 168
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Octreotide Long Acting Release | Standard Treatment
Number analyzed (Participants) | 68 | 71
Units on a scale | 0.5 (1.9) | 3.4 (2.0)

ADVERSE EVENTS:
Arm/Group | Octreotide LAR | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 15/68 | 14/71
Other Adverse Events (participants affected / at risk) | 63/68 | 68/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide LAR (N=68) | Standard Treatment (N=71)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Cardiac failure congestiv (Cardiac disorders) | 0 | 1
Diabetes mellitus (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Gastrointestinal obstruct (Gastrointestinal disorders) | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Blood alkaline phosphatas (Investigations) | 0 | 1
International normalised (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial occlusive diseas (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide LAR (N=68) | Standard Treatment (N=71)
Anaemia (Blood and lymphatic system disorders) | 15 | 11
Neutropenia (Blood and lymphatic system disorders) | 11 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 8
Diabetes mellitus (Endocrine disorders) | 4 | 3
Hypothyroidism (Endocrine disorders) | 5 | 2
Lacrimation increased (Eye disorders) | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 19 | 23
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 54 | 56
Dyspepsia (Gastrointestinal disorders) | 1 | 6
Gastritis (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 33 | 46
Vomiting (Gastrointestinal disorders) | 20 | 16
Asthenia (General disorders) | 11 | 12
Fatigue (General disorders) | 4 | 4
Mucosal inflammation (General disorders) | 7 | 3
Mucositis (General disorders) | 12 | 20
Oedema peripheral (General disorders) | 6 | 5
Pain (General disorders) | 8 | 1
Pyrexia (General disorders) | 9 | 11
Cholelithiasis (Hepatobiliary disorders) | 4 | 0
Influenza (Infections and infestations) | 6 | 11
Blood alkaline phosphatas (Investigations) | 2 | 5
Gamma-glutamyltransferase (Investigations) | 6 | 6
Weight decreased (Investigations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 17 | 14
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 11 | 12
Neuropathy peripheral (Nervous system disorders) | 18 | 21
Paraesthesia (Nervous system disorders) | 7 | 5
Anxiety (Psychiatric disorders) | 1 | 5
Insomnia (Psychiatric disorders) | 6 | 7
Dysuria (Renal and urinary disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 4
Hypertension (Vascular disorders) | 5 | 5
Hypotension (Vascular disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
Limitations were the small number of patients who received irinotecan and small proportion of patients with grade III and IV diarrhea. It is not possible to generalize our results for these populations. Study wasn't blinded or placebo-controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e. data from all sites) in the clinical trial.